CLINICAL TRIAL: NCT01894607
Title: Feasibility Study of Contrast Enhanced Intraoperative Ultrasound for Detection and Characterization of Renal Mass Undergoing Open Partial Nephrectomy
Brief Title: Contrast Enhanced Intraoperative Ultrasound for Detection and Characterization of Renal Mass Undergoing Open Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-0124; NCI-2013-02232 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Cancer
Keywords: Kidney Cancer; Renal Mass; Open partial nephrectomy; Ultrasound-guided surgery; DEFINITY; Contrast agent; Phone call
MeSH Terms: conditions — Kidney Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast Enhanced Intraoperative Ultrasound (Experimental): During standard of care surgery, radiologist will take images and videos with an ultrasound machine before patient given the contrast agent.
  Patient then receives the DEFINITY contrast by vein over about 1 minute. After receiving the injection of DEFINITY, radiologist will take more images and videos of the tumor and kidney(s) to compare to those recorded earlier.
  Follow-up phone call 30 days after standard of care surgery is complete to review any side effects patient may be having.
  Interventions: Procedure: Contrast Enhanced Intraoperative Ultrasound; Drug: DEFINITY; Behavioral: Phone Call

INTERVENTIONS:
Procedure: Contrast Enhanced Intraoperative Ultrasound — During standard of care surgery, radiologist will take images and videos with an ultrasound machine before and after patient given the contrast agent.
Drug: DEFINITY — During standard of care surgery, radiologist will take images and videos with an ultrasound machine before patient given the contrast agent.
  Patient then receives the DEFINITY contrast by vein over about 1 minute. After receiving the injection of DEFINITY, radiologist will take more images and videos of the tumor and kidney(s) to compare to those recorded earlier.
Behavioral: Phone Call — Follow-up phone call 30 days after standard of care surgery is complete to review any side effects patient may be having.

SUMMARY:
The goal of this clinical research is to learn how effective an ultrasound contrast agent, called DEFINITY, is when used during ultrasound-guided surgery to remove part of one or both kidneys.

DETAILED DESCRIPTION:
DEFINITY is a contrast agent that is used to create better quality ultrasound images.

On the day before or the day of the standard of care surgery, women who are able to become pregnant must have a negative blood or urine pregnancy test. If it a blood pregnancy test is performed, a portion of blood will be used from routine blood draws that are collected as part of your standard of care surgery.

During your standard of care surgery, the radiologist will take images and videos with an ultrasound machine before you are given the contrast agent. This is done to learn if cancer has spread around the kidney.

You will then receive the DEFINITY by vein over about 1 minute. After you receive the injection of DEFINITY, the radiologist will take more images and videos of the tumor and kidney(s) to compare to those recorded earlier.

Length of Study:

Your active participation in this study will be over after you have completed the follow-up visit.

Follow-Up Phone Call:

You will have a follow-up phone call 30 days after your standard of care surgery is complete to review any side effects you may be having. This call should take about 10 minutes to complete.

This is an investigational study. DEFINITY is FDA approved and commercially available for use in contrast enhanced echocardiography. It is not FDA approved or commercially available for use in radiology.

Up to 11 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have previous cross sectional imaging (CT or MRI) demonstrating renal mass or masses that is amenable to open partial nephrectomy.
2. Patient is scheduled for intraoperative ultrasound guided open partial nephrectomy.
3. Patient must sign informed consent, with risks and benefits of CEUS explained (see risks outlined on the following pages)

Exclusion Criteria:

1. Patients with known renal mass scheduled for total or laparoscopic partial nephrectomy.
2. Patients who are hypersensitive to Definity (Perflutren Lipid Microsphere)
3. Patients with known history of right-to-left, bidirectional or transient right-to-left cardiac shunts.
4. Pediatric patients less than 18 years of age.
5. Pregnant or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ott Le, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 07, 2013 to May 23, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Contrast Enhanced Intraoperative Ultrasound: During standard of care surgery, radiologist will take images and videos with an ultrasound machine before participant is given the contrast agent. Participant then receives the DEFINITY contrast by vein over about 1 minute. After receiving the injection of DEFINITY, radiologist will take more images and videos of the tumor and kidney(s) to compare to those recorded earlier.
Period: Overall Study
Arm/Group | Contrast Enhanced Intraoperative Ultrasound
Started | 11
Completed | 10
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Contrast Enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 52 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Successful Capture of IO-CEUS Images
Description: Primary objective is to determine feasibility of obtaining intraoperative (IO) contrast enhanced ultrasound (CEUS) images in participants undergoing open partial nephrectomy. Feasibility defined as the successful capture of IO-CEUS images in 8 out of 10 participants.
Time Frame: 1 day
Population: 1 participant was ineligible.
Measure: Number; unit: participants
Arm/Group | Contrast Enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Assess Image Quality of the Contrast Enhanced Ultrasound (CEUS)
Description: Number of participants that show better image quality in terms of lesion conspicuity and enhancement following contrast injection vs. baseline.
Time Frame: 1 day
Population: 1 participant was ineligible.
Measure: Number; unit: participants
Arm/Group | Contrast Enhanced Intraoperative Ultrasound
Number analyzed (Participants) | 10
participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were evaluated after the administration of contrast agent through the end of follow-up visit, up to 30 days.
Arm/Group | Contrast Enhanced Intraoperative Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes